CLINICAL TRIAL: NCT03633123
Title: Phase II, Multicentre, Randomized, Controlled, Two Arm, Single Blind Study to Assess Safety and Efficacy of D-PLEX Administered Concomitantly With SOC, Compared to SOC, in Prevention of Post Abdominal Surgery Incisional Infection.
Brief Title: D-PLEX 310: Safety and Efficacy of D-PLEX in the Prevention of Post Abdominal Surgery Incisional Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PolyPid Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D-PLEX 310
Record Dates: First submitted 2018-06-21; First posted 2018-08-16 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Abdominal Surgery; Colon Surgery; Post-Op Infection
Keywords: Surgical site infection; Abdominal surgery; Colon and small bowl surgery
MeSH Terms: conditions — Surgical Wound Infection | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Males and females, >18 years old, undergoing scheduled abdominal colon surgery involving resection and anastomosis or a stoma, who meet the inclusion criteria and none of the exclusion criteria and provide signed informed consent will be enrolled in the study.
  Subjects will be randomized to either the investigational arm (SOC + D-PLEX) or to the control arm (SOC only) in a 1:1 ratio.
  Subjects will be blinded to the study arm.
Who Masked: Participant
Masking Description: Subject will be blinded to the treatment arm assignment. Physicians which were not part of the team in the surgery room, or from the hospital's infectious diseases dept. will remain blinded to the study arm, and will be those assessing the incisional wound for the study primary endpoint at each follow-up visit post the index surgery.
  On top, for each suspicion of infection, an external, independent and blinded adjudication committee will be the one making the final decision whether an infection occured or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SoC) (Other): SOC prophylactic treatment pre-operation will be as per Israeli Ministry of Health and international guidelines: 1st or 2nd generation of Cephalosporine family, plus Metronidazole.
  Interventions: Other: Standard of Care (SoC)
- D-PLEX + SoC (Experimental): D-PLEX is provided to suitable and willing study subjects as an adjunct to the SoC treatment
  Interventions: Drug: D_PLEX; Other: Standard of Care (SoC)

INTERVENTIONS:
Drug: D_PLEX — D_PLEX is reconstituted into paste and administered in a single application following closure of the fascia, on the fascia suture line, and on the soft tissues of the abdominal wall along the whole length of the surgical wound (including muscle, fat and dermis).
  Arms: D-PLEX + SoC
Other: Standard of Care (SoC) — Prophylactic, pre-operation: 1st or 2nd generation of Cephalosporine family, plus Metronidazole.
  Post-operation: this is each participating center standard practice for this type of procedure

SUMMARY:
Subjects who are planned to undergo an abdominal (colon) surgery and who will meet the study entry criteria will be randomly divided into 2 groups: for half D-PLEX will be administered concomitantly with the standard of care (SOC). The other half will receive the Standard of Care treatment.

Following the surgery subjects will be followed up for additional 5 visits, at least half are in line with the routine practice of surgery Follow-Ups.

Visits will include patient safety and wound assessments.

DETAILED DESCRIPTION:
D-PLEX is a new formulation of extended controlled release of Doxycycline in the applied area for about 30 days. This study is aimed to assess the safety and efficacy of D-PLEX in prevention of post abdominal surgery incisional infection.

Eligible and willing subjects will be randomly divided, in a single-blinded manor into 2 study arms D-PLEX with SOC or SOC alone. D-PLEX will be applied during the surgery at the final stage of incision closure. All patients will be followed up for additional 5 visits over 2 months, for safety and incisional wound assessment. This will include blood tests for hematology, chemistry and PK (for some only) as well as physicians assessment of the incisional wound.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing elective abdominal colon surgery involving resection and anastomosis or a stoma.
2. Male or non-pregnant female Female of childbearing potential should have a negative serum pregnancy test prior to index procedure and agree to use a highly effective method of contraception consistently and correctly for the duration of the study.
3. Subjects who sign a written informed consent
4. Subjects who are willing and able to participate and meet all study requirements.
5. Survival expectancy of at least 60 days post randomization.

Exclusion Criteria:

1. Subjects scheduled for abdominal surgery which is classified as emergency.
2. Subjects with any preoperative active infection that is currently being treated with antibiotics.
3. Subjects receiving any antibiotic therapy in the past 4 weeks prior to enrolment besides prophylaxis or antibiotic for the treatment of the disease that consists the indication for surgery.
4. Patients undergoing concomitant additional procedures besides colon resection surgery, e.g. Hyper-thermic Intraperitoneal Chemotherapy, liver resection etc. Female sterilization surgery (i.e. salpingo-oophorectomy, hysterectomy etc.), or involvement of a small bowel procedure or Cholecystectomy may be allowed, pending an advanced consultation and approval from the sponsor.
5. Subject received chemotherapy within the last 4 weeks of surgery, or radiation for colorectal cancer to the abdomen area, prior to the planned abdominal surgery (neo- adjuvant treatment).
6. Subjects that received oral or IV doxycycline during the past 4 weeks prior to screening.
7. Subjects with known sensitivity to doxycycline and/or to the tetracycline family of drugs or to the D-PLEX's excipients.
8. Subjects with known allergies to more than 3 substances (an allergy questionnaire will be filled in during the screening process).
9. Subjects with a history of allergic/hypersensitivity reaction to any substance having required hospitalization and/or treatment with intravenous steroids/intramuscular epinephrine or in the opinion of the investigator the patient is at high risk of developing severe allergic/hypersensitivity reactions.
10. Subjects with uncontrolled Asthma (GINA III-IV).
11. Subjects with End Stage Renal Disease [Chronic Kidney Disease (CKD) stage 5].
12. Subjects with chronic urticaria.
13. Subjects diagnosed with severe neurological/cardiac events within the past 1 year prior to randomization.
14. Subjects that undergone any abdominal surgery and current planned surgery involves re-opening the scar of prior abdominal surgery.
15. Any subject with active malignancy or with malignancy that has not been in complete remission for at least 5 years.

    Excluding:
    * subjects with potentially resectable non-metastatic colorectal cancer which consists the indication for surgery. In addition,
    * patients Patients who have had carcinoma in situ of the cervix, squamous cell carcinoma of the skin and basal cell carcinoma of the skin
    * Non-violent cancer that does not require treatment 4 weeks prior to, and throughout the entire study duration will be eligible.
16. Subjects with other concurrent severe and/or uncontrolled medical condition that could compromise participation in the study (e.g. non-GI active infection, uncontrolled diabetes, uncontrolled hypertension, congestive heart failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, uncompensated cirrhosis, active upper gastrointestinal (GI) tract ulceration).
17. Psychiatric, addictive, or any other disorder that compromises ability to provide informed consent for participation in this study.
18. Chronic alcoholic or drug abuse subjects.
19. Pregnant or breast-feeding women or women of childbearing age who refuse or prohibited of using an effective contraceptive method of birth control (such as double barrier, oral or parenteral hormonal, intrauterine device and spermicide) throughout study participation including safety follow-up period.
20. Subjects that received any investigational drug within 30 days or 5½ half-lives of enrollment to the study (whichever is longer).
21. Subjects participating in any other interventional studies.
22. In the opinion of investigator, subject is not eligible to participate in the study and/or to comply with protocol requirements (e.g. due to a cognitive or medical condition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-10-06 (Actual)

PRIMARY OUTCOMES:
Infection rate as measured by the proportion of subjects with abdominal incisional infection event | By day 30 post surgery
  Infection rate as measured by the proportion of subjects with abdominal incisional infection event, as determined by a blinded and independent adjudication committee, within 30 days post abdominal surgery.

SECONDARY OUTCOMES:
Average ASEPSIS assessment score (Additional treatment, Serous discharge, Erythema, Purulent exudate, Separation of deep tissue, Isolation of bacteria, Stay duration as inpatient) during 30 days post-surgery. | At post surgery study visits : day 1, day 5, day 14 & day 30
  ASEPSIS is acronym of wound assessment and treatment parameters (described in the title), which provides numerically score during an inspection of the surgical site. The final score is being interpreted to severity of wound appearance and the clinical consequences of the infection.
  Each parameter will be evaluated and numerically scored. Some (Serous discharge & Erythema) will be marked between 0 - 5 and others (Purulent exudate & Separation of deep tissue) are marked between 0 - 10 - based on the proportion of the wound they affect when 0 is none and either 5 or 10 are for over 80% of the wound.
  Other parameters (Additional antibiotic treatment, a requirement for pus drainage, solation of bacteria & Stay duration as an inpatient) are scored Yes or No. No equals 0. Yes is calculated as either 5 points (for some parameters) or 10 for others.
  The final score can in the range of 0 - 70. 0 - 10 for wound which heals satisfactorily and over 40 for a severe wound infection.
Incidence of Deep Surgical Site Infection during 30 days post-surgery | At study visits: day 1, day 5, day 14 and day 30 post surgery
  Number of deep surgical site infections events during the 30 days post surgery, as confirmed by an independent adjudication committee.
Incidence of Superficial Surgical Site Infection during 30 days post-surgery | At study visits: day 1, day 5, day 14 and day 30 post surgery
  Number of superficial surgical site infections events during the 30 days post surgery, as confirmed by an independent adjudication committee.
Mortality rate within 60 days post abdominal surgery | During 60 days of study participation
  Death from any reason
Susceptibility to Doxycycline | At study visits: day 1, day 5, day 14 and day 30 post surgery
  Susceptibility to Doxycycline for any organisms recovered from an abdominal surgery incisional Infection site will be done using a central lab.
  When an infection is suspected in the incisional wound, a sample will be taken and sent for a bacteriology test in a central lab. Any organism which will grow (if), will be further tested for Doxycycline susceptibility.
Number of overall hospitalization days post surgery | During 60 days of study participation
  Number of hospitalization days after surgery and until discharge. Will include prolongation of primary hospitalization compared to the average of the rest of the recruited patients and re-admission due to infection
Number of re-admissions due to surgical site infection | During 60 days of study participation
  Out of the entire hospitalization period, how many days were attributed due to a surgical site infection
Number of antibiotic treatment days post surgery | During 60 days of study participation
  Number of days antibiotic treatment is administered (any route) to treat an incisional infection.
Time to surgical site infection | At study visits: day 1, day 5, day 14 and day 30 post surgery
  Number of days between surgery and a confirmed incisional surgery infection

CONTACTS AND LOCATIONS:
Overall Officials: Noam Emanuel, Dr., Study Director — Chief Scientist
Locations (8):
- Israel (8):
  - Wolfson MC, Holon
  - Meir MC, Kfar Saba
  - Rabin MC, Campus Beilinson, Petah Tikva
  - Sheba MC, Tel-Hashomer, Ramat Gan
  - Kaplan MC, Rehovot
  - Assuta Ramat-HaHayal, Tel Aviv
  - Tel-Aviv Sourasky MC, Tel Aviv
  - Assaf-Harofeh MC, Zrifin

IPD SHARING:
Plan to Share IPD: No